CLINICAL TRIAL: NCT06366282
Title: Pediatric and Caregiver Traumatic Stress Intervention: A Path Forward After Injury for Pediatric Survivors and Their Caregivers
Brief Title: Pediatric and Caregiver Traumatic Stress Intervention (PACTS)
Acronym: PACTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Childress Institute for Pediatric Trauma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00110030
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Injury
Keywords: posttraumatic stress disorder; depression; pediatric injury
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic; Depression | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peritraumatic Distress Inventory (PDI) Tool - Trauma Counseling (Experimental): Screening using Peritraumatic Distress Inventory (PDI) tool and one or more caregiver intervention during a single hospitalization
  Interventions: Behavioral: Caregiver Counseling for Childhood Traumatic Injury
- Peritraumatic Distress Inventory (PDI) Tool - Standard of Care (Active Comparator): Screening using the Peritraumatic Distress Inventory (PDI) tool and standard of care related to acute stress and post-traumatic stress
  Interventions: Behavioral: Standard of Care for Childhood Traumatic Injury

INTERVENTIONS:
Behavioral: Caregiver Counseling for Childhood Traumatic Injury — Caregiver intervention will be provided by the counseling team that includes components of trauma narrative, psychoeducation, coping strategies, and resilience-building using, for burn patients.
  Arms: Peritraumatic Distress Inventory (PDI) Tool - Trauma Counseling
Behavioral: Standard of Care for Childhood Traumatic Injury — Control group receives the current standard of care provided by the counseling team
  Arms: Peritraumatic Distress Inventory (PDI) Tool - Standard of Care

SUMMARY:
The purpose of this study is to learn more about how to help the caregiver and child survivor of a traumatic injury handle post-traumatic stress disorder and/or depression.

DETAILED DESCRIPTION:
This study is a trial to determine if a caregiver-child dyadic screening and caregiver intervention with pediatric trauma patients reduces traumatic stress symptoms in both child and caregiver, and depressive symptoms in caregivers compared to the current standard of care. The purpose of the PACTS Intervention is to identify and address the needs of the caregiver and the child survivor who are at-risk for developing post-traumatic stress disorder and/or depression following traumatic injury of the child.

ELIGIBILITY:
Inclusion Criteria:

* Child requires inpatient treatment for an unintentional injury (e.g. burns, dog bite, road traffic accident) in the pediatric trauma and/or pediatric burns units
* English-speaking adults, with English denoted as the primary language in the electronic medical record (EMR)
* Caregiver-child dyads who screen positive with the Peritraumatic Distress Inventory (PDI) Tools will be invited to participate in the randomized controlled trial.

Exclusion Criteria:

* Patients and/or caregivers with cognitive deficits, with psychotic symptoms, refusing treatment, and leaving the hospital against medical advice (AMA) were unable to participate in counseling interventions by condition or by choice and are excluded from the study population

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Kessler 6 Scores | From baseline to Month 3
  Administered to the caregiver to screen for secondary Post Traumatic Stress Disorder (PTSD) - A six-item K6 screening scale for psychological distress - a short measure of non-specific psychological distress based on questions about the level of nervousness, agitation, psychological fatigue and depression - scores range from 10-50 with higher scores meaning a severe mental disorder
Change in Patient Health Questionnaire - 9 (PHQ-9) Scores | From baseline to Month 3
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression
Change in Child and Adolescent Trauma Screen (CATS) Scores | From baseline to Month 3
  Caregiver administered to caregiver to screen for PTSD in the child - The "Child and Adolescent Trauma Screen (CATS)" is a Diagnostic and Statistical Manual-5 (DSM-5) based checklist that includes 15 potentially traumatic events or series of events, the 20 posttraumatic stress symptoms (PTSS) and 5 impairment items. The younger child version conforms to the DSM-5 3-6 year old PTSD symptom criteria. The CATS can be administered as a self-report or as an interview. Interview may be preferable with younger children or youth with reading comprehension challenges. Scores ranging from 0-16+ with higher scores meaning more probability of Post Traumatic Stress Disorder (PTSD)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shilling, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No